CLINICAL TRIAL: NCT04089423
Title: Prospective Multicentre Evaluation of the Accuracy and Diagnostic Yield of the Fujifilm SILVAMP TB LAM (FujiLAM) Test for the Diagnosis of Tuberculosis in People Living With HIV
Brief Title: FujiLAM Prospective Evaluation Trial
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); Infectious Diseases Institute, Uganda (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); Swiss Tropical & Public Health Institute (Other); Ifakara Health Institute (Other); University of Cape Town (Other); Viet Tiep Hospital (Other); National Tuberculosis Control Programme (Unknown); Fujifilm (Industry); Omega Diagnostics (Unknown); Tuberculosis and Lung Disease Hospital in Hai Phong (Unknown); The HIV Netherlands Australia Thailand Research Collaboration (Other)
Responsible Party: Sponsor
Other Study IDs: 7430-2/1
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Diagnosis of Tuberculosis in People Living With HIV
Keywords: tuberculosis, PLHIV
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fujifilm SILVAMP TB LAM — Fujifilm SILVAMP TB LAM detects the presence of lipoarabinomannan (LAM) in urine with a visually read lateral flow test that uses silver amplification.
  Other Names: Omega VISITECT® CD4 Advanced Disease test

SUMMARY:
This is a prospective, multicentre cohort study in which the accuracy and the diagnostic yield of the FujiLAM test will be assessed using a microbiological reference standard, an extended microbiological reference standard and a composite reference standard among inpatient and outpatient people living with HIV (PLHIV).

ELIGIBILITY:
Inclusion Criteria:

* Adult PLHIV (≥18 years), irrespective of their CD4 count and antiretroviral therapy (ART) status, at risk of having pulmonary and/or extra-pulmonary TB
* Inpatients: irrespective of TB symptoms
* Outpatients: at least one of the symptoms suggestive of TB (as defined by WHO*)
* written informed consent
* willingness to have a trial follow-up visit at 2-3 and 6 months after enrolment (e.g. not planning to relocate)

Exclusion Criteria:

* Current anti-TB treatment *
* Any anti-TB treatment within 60 days prior to enrolment
* Any isoniazid preventive therapy within 6 months prior to enrolment * Patients starting anti-TB treatment at the time of enrolment will not be excluded from the trial provided that all trial specimens are collected before starting the 3rd dose of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult people living with HIV
Sampling Method: Probability Sample
Enrollment: 1731 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Point estimates of sensitivity and specificity of FujiLAM, with 95% confidence intervals, using the defined eMRS. | Day 1
Point estimates of sensitivity and specificity of FujiLAM, with 95% confidence intervals, using the defined CRS. | Day 1
Diagnostic yield, with 95% confidence interval, of FujiLAM test among eMRS positive patients and AlereLAM, Smear and Ultra (sputum, urine) as comparators (on Day 1 specimens). | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Morten Ruhwald, MD, Principal Investigator — FIND Head of TB programme
Locations (7):
- Malawi-Liverpool-Wellcome Trust Clinical Research Programme, Blantyre, Malawi
- CIDRI-Africa University of Cape Town, Cape Town, South Africa
- Ifakara Health Institute, Dar es Salaam, Tanzania
- The HIV Netherlands Australia Thailand Research collaboration, Bangkok, Bankok, Thailand
- Infectious Diseases Institute, Kampala, Uganda
- Viet Tiep Hospital, Haiphong, Le Chan, Vietnam
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sossen B, Szekely R, Mukoka M, Muyoyeta M, Nakabugo E, Hella J, Van Nguyen H, Ubolyam S, Erkosar B, Vermeulen M, Centner CM, Nyangu S, Sanjase N, Sasamalo M, Dinh HT, Ngo TA, Manosuthi W, Jirajariyavej S, Nguyen NV, Avihingsanon A, Kerkhoff AD, Denkinger CM, Reither K, Nakiyingi L, MacPherson P, Meintjes G, Ruhwald M; FujiLAM Study Consortium. Urine-Xpert Ultra for the diagnosis of tuberculosis in people living with HIV: a prospective, multicentre, diagnostic accuracy study. Lancet Glob Health. 2024 Dec;12(12):e2024-2034. doi: 10.1016/S2214-109X(24)00357-7. PMID 39577975
- [Derived] Gils T, Hella J, Jacobs BKM, Sossen B, Mukoka M, Muyoyeta M, Nakabugo E, Van Nguyen H, Ubolyam S, Mace A, Vermeulen M, Nyangu S, Sanjase N, Sasamalo M, Dinh HT, Ngo TA, Manosuthi W, Jirajariyavej S, Denkinger CM, Nguyen NV, Avihingsanon A, Nakiyingi L, Szekely R, Kerkhoff AD, MacPherson P, Meintjes G, Reither K, Ruhwald M. A Prospective Evaluation of the Diagnostic Accuracy of the Point-of-Care VISITECT CD4 Advanced Disease Test in 7 Countries. J Infect Dis. 2025 Feb 4;231(1):e82-e90. doi: 10.1093/infdis/jiae374. PMID 39046150
- [Derived] Szekely R, Sossen B, Mukoka M, Muyoyeta M, Nakabugo E, Hella J, Nguyen HV, Ubolyam S, Chikamatsu K, Mace A, Vermeulen M, Centner CM, Nyangu S, Sanjase N, Sasamalo M, Dinh HT, Ngo TA, Manosuthi W, Jirajariyavej S, Mitarai S, Nguyen NV, Avihingsanon A, Reither K, Nakiyingi L, Kerkhoff AD, MacPherson P, Meintjes G, Denkinger CM, Ruhwald M; FujiLAM Study Consortium. Prospective multicentre accuracy evaluation of the FUJIFILM SILVAMP TB LAM test for the diagnosis of tuberculosis in people living with HIV demonstrates lot-to-lot variability. PLoS One. 2024 May 31;19(5):e0303846. doi: 10.1371/journal.pone.0303846. eCollection 2024. PMID 38820372